CLINICAL TRIAL: NCT00242567
Title: A Phase III, Parallel Group, Randomized, Open-label, Multi-centre Clinical Trial of Zoledronic Acid in Males Receiving Androgen Deprivation Therapy for Advanced Prostate Cancer.
Brief Title: Study of Zoledronic Acid for Patients With Hormone-sensitive Bone Metastases From Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446E2432
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Prostate Cancer
Keywords: zoledronic acid; bone metastases; prostate cancer; hormone-sensitive
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid; Androgen Antagonists

ARMS (2):
- Early Group (Experimental): Zoledronic acid 4 mg i.v. infusion every 4 weeks, commencing at Baseline.
  Interventions: Drug: Zoledronic Acid
- Delayed group (Experimental): Zoledronic acid 4 mg i.v. infusion every 4 weeks, commencing no sooner than 12 months after their baseline visit, and not until they have had three rises in PSA level from Baseline, one of which must be a least 10 ng/mL greater than the baseline Serum Prostate-specific Antigen (PSA) level.
  Interventions: Drug: Androgen Deprivation Therapy (ADT)

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid was provided by Novartis in vials containing 4 mg/5 mL liquid concentrate. Prior to administration, the liquid concentrate from one vial was to be further diluted with 100 mL of calcium-free infusion solution (0.9 % weight by volume sodium chloride solution or 5 % weight by volume glucose solution). If refrigerated, the solution had to be allowed to reach room temperature before administration.
  After addition of the liquid concentrate to the infusion media, the infusion solution was to be used as soon as practicable to reduce the risk of microbiological hazard. If storage of the solution was necessary, it had to be refrigerated at temperatures between 2-8 degrees C and was to be used within 24 hours.
  The infusion solution containing 4 mg zoledronic acid was to be administered every 4 weeks as an i.v. infusion over no less than 15 minutes.
  Arms: Early Group
Drug: Androgen Deprivation Therapy (ADT) — Androgen deprivation therapy (ADT) was to be administered according to institutional protocols, in accordance with relevant prescribing information. The type and duration of androgen deprivation was at the discretion of the treating specialist, and could include orchiectomy where this would normally have been performed. Androgen deprivation therapy was provided by the investigational center, or obtained by the patient from usual sources. Anti-androgen monotherapy and intermittent ADT were excluded in the first 12 months of the study.
  Arms: Delayed group

SUMMARY:
This study aims to determine whether early treatment with zoledronic acid, that is given during the early phase of advanced prostate cancer, will be more efficacious than delayed treatment

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer
* at least one bone metastasis
* receiving or about to receive androgen deprivation therapy (ADT)

Exclusion Criteria:

* previous ADT failure
* previous or current treatment with another bone-protecting agent, chemotherapy or targeted therapy
* abnormal renal function

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2005-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- Australia (5):
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Brisbane
  - Novartis Investigative Site, Melbourne
  - Novartis Investigative Site, Port Macquarie
  - Novartis Investigative Site, Sydney
- Brazil (3):
  - Novartis Investigative Site, Porto Alegre
  - Novartis Investigative Site, Santo André
  - Novartis Investigative Site, São Paulo
- China (3):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Kuwait City, Kuwait
- Novartis Investigative Site, Beirut, Lebanon
- New Zealand (5):
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Hamilton
  - Novartis Investigative Site, Tauranga
  - Novartis Investigative Site, Wellington
- Novartis Investigative Site, Riyadh, Saudi Arabia
- South Korea (3):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Kyunggi-do
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Songkhla

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 552 patients enrolled, but 30 patients were excluded due to GCP issues in one country.
Groups:
- Delayed Group: Zoledronic acid 4 mg i.v. infusion every 4 weeks, commencing no sooner than 12 months after their baseline visit, and not until they have had three rises in PSA level from Baseline, one of which must be a least 10 ng/mL greater than the baseline PSA level.
Period: Overall Study
Arm/Group | Early Group | Delayed Group
Started | 259 | 263
Received at Least 1 Dose of Study Drug | 259 | 72
Never Received Study Drug | 0 | 191
Completed | 93 | 123
Not Completed | 166 | 140
Not completed — Adverse Event | 70 | 43
Not completed — Disease Progression | 17 | 22
Not completed — Symptomatic deterioration | 9 | 3
Not completed — Lack of Efficacy | 2 | 2
Not completed — Lost to Follow-up | 9 | 19
Not completed — Withdrawal by Subject | 33 | 28
Not completed — Protocol Violation | 12 | 12
Not completed — Use of an inhibitor of bone resorption | 0 | 2
Not completed — Other | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Group | Delayed Group | Total
Number analyzed (Participants) | 259 | 263 | 522
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (8.46) | 70.2 (8.26) | 69.8 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 259 | 263 | 522

OUTCOME MEASURES:

1. Primary Outcome: Skeletal-related Event-free Survival in Men With Bone Metastases From Prostate Cancer
Description: Skeletal-related event free survival is the time from randomization until the first detected Skeletal Related Event (SRE). Patients who were still SRE-free at 18 months were censored.
Time Frame: 18 months
Population: The ITT Population will consist of all patients randomized to treatment.
Measure: Number; unit: participants
Arm/Group | Early Group | Delayed Group
Number analyzed (Participants) | 259 | 263
participants
  Patients with event (s) | 58 | 49
  Patients without event (censored) | 201 | 214

2. Secondary Outcome: Overall Survival at 18 Months and 3 Years
Description: Overall survival (OS) time was measured from the start of study drug to the date of death due to any cause.
Time Frame: month 18, year 3
Population: The ITT Population will consist of all patients randomized to treatment.
Measure: Number; unit: participants
Arm/Group | Early Group | Delayed Group
Number analyzed (Participants) | 259 | 263
participants
  Patients with event (s) - 18 months | 31 | 21
  Patients without event - 18 months | 228 | 242
  Patients with event (s) - 36 months | 49 | 44
  Patients without event - 36 months | 210 | 219

3. Secondary Outcome: Time to Occurrence of Skeletal Related Event or Death
Description: Time from randomization to the first detected skeletal related event or death. This endpoint is the same as the primary endpoint with the modification that deaths are considered events.
Time Frame: 18 Months
Population: The ITT Population consisted of all patients randomized to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Early Group | Delayed Group
Number analyzed (Participants) | 259 | 263
Days | NA [NA to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE or Death at 18 months | NA [NA to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE or Death at 18 months

4. Secondary Outcome: Skeletal-related Event(SRE)-Free Survival
Description: Time from randomization until the first detected SRE. Patients who were still SRE-free at 3 years were censored.
Time Frame: 36 months
Population: The ITT Population consisted of all patients randomized to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Early Group | Delayed Group
Number analyzed (Participants) | 259 | 263
Days | NA [NA to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE at 36 months | NA [NA to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE at 36 months

5. Secondary Outcome: Time to Occurrence of Skeletal Related Event or Death
Description: as for outcome 3
Time Frame: 36 Months
Population: The ITT Population consisted of all patients randomized to treatment.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Early Group | Delayed Group
Number analyzed (Participants) | 259 | 263
Days | NA [945 to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE or Death at 36 months | NA [NA to NA] — Median time to event was not calculable due to less than 50% of patients had an event of SRE or Death at 36 months

ADVERSE EVENTS:
Groups:
- Early Group: Early Group
- Delayed Group (Overall): Delayed Group (Overall)
- Delayed Group (No Zometa): Delayed Group (No Zometa)
- Delayed Group (Zometa): Delayed Group (Zometa)
Arm/Group | Early Group | Delayed Group (Overall) | Delayed Group (No Zometa) | Delayed Group (Zometa)
Serious Adverse Events (participants affected / at risk) | 121/259 | 104/263 | 67/191 | 37/72
Other Adverse Events (participants affected / at risk) | 220/259 | 197/263 | 135/191 | 62/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Group (N=259) | Delayed Group (Overall) (N=263) | Delayed Group (No Zometa) (N=191) | Delayed Group (Zometa) (N=72)
ANAEMIA (Blood and lymphatic system disorders) | 7 | 11 | 7 | 4
BONE MARROW FAILURE (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
PROTEIN DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 1 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 1 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 3 | 2 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 3 | 2 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 | 1 | 1 | 0
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 1 | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 2 | 3 | 3 | 0
CARDIAC DISCOMFORT (Cardiac disorders) | 0 | 1 | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 1 | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 | 0 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 3 | 1 | 2
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 3 | 0 | 0 | 0
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 1 | 1 | 0
CARDIOTOXICITY (Cardiac disorders) | 0 | 1 | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 1 | 0 | 1
CORONARY ARTERY STENOSIS (Cardiac disorders) | 1 | 0 | 0 | 0
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 | 0 | 0 | 0
LEFT VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 | 1 | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 2 | 2 | 0
PALPITATIONS (Cardiac disorders) | 0 | 1 | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0
PHIMOSIS (Congenital, familial and genetic disorders) | 0 | 1 | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
GOITRE (Endocrine disorders) | 0 | 1 | 1 | 0
CATARACT (Eye disorders) | 2 | 1 | 1 | 0
CATARACT NUCLEAR (Eye disorders) | 1 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 1 | 0 | 0 | 0
EYE PAIN (Eye disorders) | 1 | 0 | 0 | 0
OPHTHALMOPLEGIA (Eye disorders) | 1 | 0 | 0 | 0
ORBITAL OEDEMA (Eye disorders) | 1 | 0 | 0 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0 | 0 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0 | 0
VISUAL IMPAIRMENT (Eye disorders) | 1 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1 | 0 | 1
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1
CAECITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 3 | 1 | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 3 | 2 | 1
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1
DUODENAL ULCER PERFORATION (Gastrointestinal disorders) | 1 | 1 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0 | 1
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 1 | 0 | 1
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 0 | 1 | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 2 | 1 | 1
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PEPTIC ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0
PROCTITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 1
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 2 | 2 | 0
VOMITING (Gastrointestinal disorders) | 7 | 2 | 1 | 1
ABASIA (General disorders) | 0 | 1 | 1 | 0
ASTHENIA (General disorders) | 5 | 6 | 4 | 2
CATHETER SITE PAIN (General disorders) | 0 | 1 | 1 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0 | 0
CHEST PAIN (General disorders) | 2 | 2 | 1 | 1
CHILLS (General disorders) | 0 | 1 | 1 | 0
CONCOMITANT DISEASE PROGRESSION (General disorders) | 2 | 3 | 3 | 0
DEATH (General disorders) | 4 | 5 | 2 | 3
DISEASE PROGRESSION (General disorders) | 25 | 16 | 10 | 6
DRUG INEFFECTIVE (General disorders) | 1 | 0 | 0 | 0
FACE OEDEMA (General disorders) | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 1 | 4 | 4 | 0
FEELING COLD (General disorders) | 1 | 0 | 0 | 0
GAIT DISTURBANCE (General disorders) | 2 | 1 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 1 | 0 | 1
GENERALISED OEDEMA (General disorders) | 0 | 1 | 1 | 0
MALAISE (General disorders) | 1 | 0 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0 | 0 | 0
MULTI-ORGAN DISORDER (General disorders) | 1 | 1 | 0 | 1
MULTI-ORGAN FAILURE (General disorders) | 4 | 1 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 3 | 1 | 2
PAIN (General disorders) | 2 | 1 | 1 | 0
PELVIC MASS (General disorders) | 0 | 1 | 0 | 1
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 0 | 0 | 0
PYREXIA (General disorders) | 6 | 0 | 0 | 0
SUPRAPUBIC PAIN (General disorders) | 1 | 0 | 0 | 0
ULCER (General disorders) | 0 | 1 | 1 | 0
BILIARY DILATATION (Hepatobiliary disorders) | 1 | 0 | 0 | 0
BUDD-CHIARI SYNDROME (Hepatobiliary disorders) | 0 | 1 | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 2 | 2 | 0
HEPATIC INFARCTION (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HEPATIC LESION (Hepatobiliary disorders) | 1 | 0 | 0 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 0 | 1 | 1 | 0
HEPATOMEGALY (Hepatobiliary disorders) | 0 | 1 | 0 | 1
HEPATORENAL FAILURE (Hepatobiliary disorders) | 2 | 1 | 1 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 1 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 0 | 1 | 0 | 1
ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 1 | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 2 | 4 | 1 | 3
CARBUNCLE (Infections and infestations) | 0 | 1 | 1 | 0
CELLULITIS (Infections and infestations) | 2 | 0 | 0 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 1 | 0 | 1
DIVERTICULITIS (Infections and infestations) | 2 | 0 | 0 | 0
ECZEMA INFECTED (Infections and infestations) | 0 | 1 | 0 | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0 | 0 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 4 | 2 | 2 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1 | 0 | 1
INFECTED SKIN ULCER (Infections and infestations) | 0 | 1 | 1 | 0
INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
INFLUENZA (Infections and infestations) | 2 | 0 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 3 | 3 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 1 | 0
LUNG INFECTION (Infections and infestations) | 1 | 1 | 0 | 1
NECROTISING FASCIITIS (Infections and infestations) | 0 | 1 | 1 | 0
NOSOCOMIAL INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 0
OROPHARYNGITIS FUNGAL (Infections and infestations) | 1 | 0 | 0 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0 | 0 | 0
OSTEOMYELITIS CHRONIC (Infections and infestations) | 1 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 8 | 3 | 2 | 1
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 1 | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
RECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
SEPSIS (Infections and infestations) | 4 | 5 | 5 | 0
SEPTIC SHOCK (Infections and infestations) | 2 | 1 | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 7 | 6 | 5 | 1
UROSEPSIS (Infections and infestations) | 0 | 1 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
WOUND INFECTION (Infections and infestations) | 0 | 1 | 1 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 3 | 2 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
GASTROENTERITIS RADIATION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
PENIS INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
SKELETAL INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 3 | 3 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 0 | 1 | 0 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD CREATINE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD CREATININE (Investigations) | 0 | 1 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 3 | 2 | 2 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD MAGNESIUM INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD PHOSPHORUS INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD POTASSIUM INCREASED (Investigations) | 1 | 0 | 0 | 0
BLOOD TESTOSTERONE INCREASED (Investigations) | 0 | 2 | 0 | 2
BONE SCAN ABNORMAL (Investigations) | 1 | 0 | 0 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0 | 0 | 0
ELECTROCARDIOGRAM ST-T CHANGE (Investigations) | 1 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 2 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0 | 0
HEPATITIS C POSITIVE (Investigations) | 0 | 1 | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1 | 0 | 1
LYMPHOCYTE COUNT DECREASED (Investigations) | 0 | 1 | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 0 | 2 | 1 | 1
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 0 | 3 | 2 | 1
PROTEIN TOTAL DECREASED (Investigations) | 0 | 1 | 0 | 1
TROPONIN INCREASED (Investigations) | 1 | 0 | 0 | 0
URINE OUTPUT DECREASED (Investigations) | 2 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 2 | 1 | 1 | 0
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 4 | 4 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 2 | 2 | 0
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
FLUID INTAKE REDUCED (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
HYPOPHAGIA (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
MARASMUS (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 6 | 2 | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
BONE MARROW TUMOUR CELL INFILTRATION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
BONE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
HEAD AND NECK CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 1 | 1
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 1 | 4
METASTASES TO BONE MARROW (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 0 | 2
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 1
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 1
METASTASES TO LYMPH NODES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
METASTASES TO NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
NEUROENDOCRINE TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
ORAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
PANCOAST'S TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 22 | 13 | 9
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8 | 5 | 3
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 2 | 1 | 1 | 0
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 1
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 0 | 1 | 0 | 1
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 1 | 0
CAUDA EQUINA SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 1
CEREBELLAR INFARCTION (Nervous system disorders) | 0 | 1 | 0 | 1
CEREBRAL ARTERY OCCLUSION (Nervous system disorders) | 0 | 1 | 0 | 1
CEREBRAL ARTERY STENOSIS (Nervous system disorders) | 0 | 1 | 0 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 4 | 4 | 4 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 3 | 2 | 0 | 2
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 3 | 2 | 1
COMA HEPATIC (Nervous system disorders) | 1 | 0 | 0 | 0
COMA URAEMIC (Nervous system disorders) | 0 | 1 | 1 | 0
CONVULSION (Nervous system disorders) | 1 | 2 | 1 | 1
DEMENTIA (Nervous system disorders) | 1 | 0 | 0 | 0
DIABETIC MONONEUROPATHY (Nervous system disorders) | 0 | 1 | 1 | 0
DYSSTASIA (Nervous system disorders) | 1 | 0 | 0 | 0
FACIAL PALSY (Nervous system disorders) | 0 | 1 | 0 | 1
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 2 | 2 | 0
HORNER'S SYNDROME (Nervous system disorders) | 1 | 0 | 0 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 0 | 0
HYPOGLYCAEMIC COMA (Nervous system disorders) | 0 | 1 | 1 | 0
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 1 | 0 | 0 | 0
LACUNAR INFARCTION (Nervous system disorders) | 1 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1 | 1 | 0
PARAPARESIS (Nervous system disorders) | 1 | 0 | 0 | 0
PARAPLEGIA (Nervous system disorders) | 1 | 2 | 1 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 6 | 3 | 3 | 0
SPINAL MENINGEAL CYST (Nervous system disorders) | 1 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 3 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 1 | 0 | 1
ANXIETY (Psychiatric disorders) | 1 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1 | 0
DISORIENTATION (Psychiatric disorders) | 1 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1 | 1 | 0
ANURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0
AZOTAEMIA (Renal and urinary disorders) | 0 | 1 | 1 | 0
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 | 1 | 0 | 1
BLADDER OBSTRUCTION (Renal and urinary disorders) | 1 | 0 | 0 | 0
CALCULUS BLADDER (Renal and urinary disorders) | 0 | 1 | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0 | 0 | 0
DYSURIA (Renal and urinary disorders) | 3 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 3 | 3 | 0 | 3
HYDRONEPHROSIS (Renal and urinary disorders) | 4 | 1 | 0 | 1
NOCTURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0
POLYURIA (Renal and urinary disorders) | 0 | 1 | 1 | 0
PYELOCALIECTASIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 5 | 1 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 5 | 4 | 4 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 | 2 | 2 | 0
RENAL INFARCT (Renal and urinary disorders) | 1 | 0 | 0 | 0
URETERAL DISORDER (Renal and urinary disorders) | 0 | 1 | 0 | 1
URETERIC OBSTRUCTION (Renal and urinary disorders) | 2 | 0 | 0 | 0
URETHRAL DILATATION (Renal and urinary disorders) | 1 | 0 | 0 | 0
URETHRAL STENOSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 1 | 1 | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 1 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 5 | 6 | 3 | 3
URINARY TRACT DISORDER (Renal and urinary disorders) | 0 | 1 | 0 | 1
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 | 2 | 2 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 2 | 2 | 0
BREAST PAIN (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PENILE PAIN (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 | 1 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1 | 1
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 1 | 0 | 0 | 0
AORTIC ANEURYSM (Vascular disorders) | 1 | 0 | 0 | 0
ARTERIAL STENOSIS LIMB (Vascular disorders) | 1 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 2 | 0 | 2
EXTRINSIC VASCULAR COMPRESSION (Vascular disorders) | 0 | 1 | 0 | 1
HAEMORRHAGE (Vascular disorders) | 0 | 1 | 1 | 0
HYPERTENSION (Vascular disorders) | 4 | 0 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0 | 0 | 0
SHOCK (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Early Group (N=259) | Delayed Group (Overall) (N=263) | Delayed Group (No Zometa) (N=191) | Delayed Group (Zometa) (N=72)
ANAEMIA (Blood and lymphatic system disorders) | 39 | 30 | 12 | 18
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 6 | 1 | 5
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 4 | 0 | 4
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 10 | 6 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 | 14 | 9 | 5
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 13 | 4 | 2 | 2
CONSTIPATION (Gastrointestinal disorders) | 46 | 53 | 33 | 20
DIARRHOEA (Gastrointestinal disorders) | 27 | 23 | 17 | 6
DYSPEPSIA (Gastrointestinal disorders) | 11 | 7 | 3 | 4
NAUSEA (Gastrointestinal disorders) | 30 | 28 | 14 | 14
VOMITING (Gastrointestinal disorders) | 23 | 12 | 6 | 6
ASTHENIA (General disorders) | 17 | 13 | 6 | 7
FATIGUE (General disorders) | 31 | 21 | 9 | 12
INFLUENZA LIKE ILLNESS (General disorders) | 28 | 12 | 6 | 6
OEDEMA PERIPHERAL (General disorders) | 29 | 23 | 14 | 9
PAIN (General disorders) | 15 | 12 | 8 | 4
PYREXIA (General disorders) | 30 | 8 | 3 | 5
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 14 | 11 | 3
NASOPHARYNGITIS (Infections and infestations) | 19 | 17 | 11 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 28 | 20 | 14 | 6
URINARY TRACT INFECTION (Infections and infestations) | 15 | 22 | 13 | 9
FALL (Injury, poisoning and procedural complications) | 16 | 17 | 11 | 6
SKIN LACERATION (Injury, poisoning and procedural complications) | 3 | 10 | 6 | 4
BLOOD CREATININE INCREASED (Investigations) | 56 | 27 | 18 | 9
PROSTATIC SPECIFIC ANTIGEN INCREASED (Investigations) | 60 | 61 | 26 | 35
WEIGHT DECREASED (Investigations) | 15 | 19 | 12 | 7
WEIGHT INCREASED (Investigations) | 7 | 10 | 6 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 35 | 24 | 12 | 12
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 33 | 11 | 4 | 7
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 15 | 6 | 1 | 5
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 53 | 46 | 28 | 18
BACK PAIN (Musculoskeletal and connective tissue disorders) | 61 | 54 | 28 | 26
BONE PAIN (Musculoskeletal and connective tissue disorders) | 34 | 30 | 18 | 12
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 15 | 6 | 3 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 10 | 14 | 7 | 7
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 9 | 20 | 12 | 8
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 6 | 8 | 3 | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 31 | 26 | 17 | 9
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 6 | 7 | 2 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 18 | 15 | 9 | 6
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 7 | 2 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 36 | 42 | 18 | 24
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 11 | 7 | 4
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 13 | 4 | 9
DIZZINESS (Nervous system disorders) | 18 | 17 | 11 | 6
HEADACHE (Nervous system disorders) | 19 | 8 | 5 | 3
HYPOAESTHESIA (Nervous system disorders) | 9 | 5 | 1 | 4
PARAESTHESIA (Nervous system disorders) | 16 | 9 | 5 | 4
DEPRESSED MOOD (Psychiatric disorders) | 4 | 4 | 0 | 4
INSOMNIA (Psychiatric disorders) | 19 | 18 | 9 | 9
DYSURIA (Renal and urinary disorders) | 17 | 15 | 9 | 6
HAEMATURIA (Renal and urinary disorders) | 17 | 11 | 5 | 6
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 5 | 1 | 4
NOCTURIA (Renal and urinary disorders) | 16 | 13 | 5 | 8
POLLAKIURIA (Renal and urinary disorders) | 10 | 9 | 5 | 4
URINARY RETENTION (Renal and urinary disorders) | 9 | 7 | 2 | 5
PELVIC PAIN (Reproductive system and breast disorders) | 7 | 7 | 2 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 | 17 | 12 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 | 18 | 9 | 9
HOT FLUSH (Vascular disorders) | 18 | 24 | 15 | 9
HYPERTENSION (Vascular disorders) | 14 | 11 | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators are NOT employed by the organization sponsoring the study. Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed.

The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial.